CLINICAL TRIAL: NCT00138320
Title: Transfer of Herpes Simplex Virus Type 2 gD Subunit Vaccine-Induced Antibodies From Mothers to Neonates
Brief Title: Herpevac Neonatal Substudy
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 04-041
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-08

CONDITIONS: Herpes Simplex
Keywords: Herpes Simplex, vaccine, antibodies, mother
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera obtained from collected blood samples will be used. Ten mL of blood will be collected at the maternal blood draw and from the umbilical vein. Three to 5 mL of blood will be collected at each infant blood draw

SUMMARY:
The purpose of this study to look at the antibodies (proteins from the body's infection fighting system) in the blood of babies delivered by women who are participants in the Herpevac Trial for Women, and who were vaccinated with either two or three doses of (GlaxoSmithKline) GSK candidate vaccine gD2t/alum-MPL or hepatitis A vaccine. The goal of this study is to compare the herpes or hepatitis A antibody levels of the newborns to those of their mothers, and to see how much of the antibodies are still present in the baby at two and six months after birth. Approximately 2 teaspoons (10 ml) of the mother's blood will be collected at the time of delivery or within 15 days before or after delivery. Approximately 2 teaspoons of blood will be collected from the child's umbilical cord at the time of delivery, or 1 teaspoon (3-5 ml) of the child's blood will be drawn within 15 days after birth. Optional blood draws from babies may occur 2 and 6 months after birth.

DETAILED DESCRIPTION:
The primary objective of this study is to quantitate HSV-2 binding and neutralizing antibody titers in the sera of newborns delivered by HSV-uninfected women vaccinated with either two or three doses of GSK candidate vaccine gD2t/alum-MPL and to compare the HSV-2 binding and neutralizing antibody titers of the newborns to those of their mothers. Secondary objectives are to: 1) evaluate the durability of HSV-2 binding and neutralizing antibody titers in the sera of newborns delivered by HSV-uninfected women vaccinated with either two or three doses of GSK candidate vaccine gD2t/alum-MPL; and 2) quantitate hepatitis A binding antibody titers in the sera of newborns delivered by women vaccinated with either two or three doses of Havrix® hepatitis A vaccine (the control vaccine used in the Herpevac Trial for Women), compare hepatitis A binding antibody titers of the newborns to those of their mothers, and evaluate the durability of hepatitis A binding antibodies in these newborns. The sample size for this study cannot be determined but based on experience is not likely to be more than 50 women. Optional additional blood will be collected from the mother and her infant at 2 mos and 6 mos after delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the Herpevac Trial for Women.
2. Has received at least two doses of either the candidate or control vaccine.
3. Pregnant.
4. Written informed consent obtained from the participant.
5. Willing to have her blood collected either at the time of delivery or within 15 days before or after delivery. If blood is to be collected by the health care provider who will be presiding at the delivery, the participant must be willing to give permission for study personnel to contact that health care provider to arrange the collection of blood.
6. Willing to have either umbilical vein blood collected at the time of delivery or blood collected from her neonate within 15 days after delivery. If blood is to be collected from the umbilical vein, the participant must be willing to give permission for study personnel to contact the presiding health care provider to arrange the collection of blood.
7. A participant whom the investigator believes can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. Termination of the pregnancy, other than live birth.
2. Entry violation in the Herpevac Trial for Women at enrollment.
3. Receipt of immunoglobulin or blood products within 4 months prior to expected date of delivery.
4. History or current clinical evidence of herpes simplex virus infection.

Maternal withdrawal criteria: If any of the following occur after enrollment, the subject will be withdrawn prior to obtaining any blood samples:

1. Termination of the pregnancy, other than live birth.
2. Determination that the subject was enrolled in the Herpevac Trial for Women in violation of that study's entry criteria.
3. Receipt of immunoglobulin or blood products within 4 months prior to expected or actual date of delivery.
4. Inability to collect umbilical vein blood at the time of delivery or neonatal blood within 15 days after birth due to logistical or other reasons.

Infant withdrawal criteria: If any of the following occurs during the study, the 2 and 6-month blood samples (or the 6-month sample only if the occurrence follows the 2-month blood draw) will not be collected from the infant:

1. Participant [mother] chooses not to participate, or continue her participation in, the optional arm of the study.
2. Inability to collect neonatal blood within 15 days after birth due to logistical or other reasons from infants for whom umbilical vein blood was not collected.
3. Death of the infant.
4. Adoption of the infant prior to completion of the study.
5. At the discretion of the investigator.
6. Receipt of immunoglobulin or blood products by the infant prior to blood draw.

Max Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who become pregnant while enrolled as participants in the Herpevac Trial for Women, DMID Protocol 01-643
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah